CLINICAL TRIAL: NCT02864017
Title: Immuno Nutrition by L-citrulline for Critically Ill Patients
Acronym: Immunocitre
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 35RC14_9835; 2015-A00961-48 (Other: Id-RCB)
Record Dates: First submitted 2016-08-04; First posted 2016-08-11 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Intubation; Pulmonary Ventilation
MeSH Terms: interventions — Enteral Nutrition; Citrulline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-Citrulline group (Experimental): Enteral nutrition 5-day L-citrulline treatment (10 grams/day)
  Interventions: Procedure: Enteral nutrition; Dietary Supplement: L-Citrulline
- Control group (Placebo Comparator): Enteral nutrition 5-day placebo treatment
  Interventions: Procedure: Enteral nutrition; Dietary Supplement: Placebo

INTERVENTIONS:
Procedure: Enteral nutrition
Dietary Supplement: L-Citrulline
  Arms: L-Citrulline group
Dietary Supplement: Placebo
  Arms: Control group

SUMMARY:
The main objective of this study is to demonstrate that the only administration of L-citrulline, can improve immune functions in critically ill patients at high risk of nosocomial infection.

DETAILED DESCRIPTION:
This is a multicentric therapeutic trial, randomized and double blind: standard enteral nutrition plus L-citrulline (5 grams/12 Hours for 5 days from the admission in Intensive Care Unit (ICU)) versus standard enteral nutrition plus placebo.

Methods-Patients: Non-surgical patients admitted in medical intensive care unit, under mechanical ventilation for an expected duration > 2 days, without severe sepsis or septic shock, will be enrolled. Symptoms leading for ICU admission ongoing for five days maximum. On admission (before treatment), the severity will be evaluated with the Sepsis-related Organ Failure Assessment (SOFA) score together with an assessment of plasmatic arginine, cytokines (InterLeukin-6 (IL6) ), and expression of Human Leukocyte Antigen - antigen D Related (HLA-DR) by monocytes. The same evaluation will be repeated on day 3 (during treatment) and on day 7 (after treatment).

The enrolment of 100 patients is statistically enough to demonstrate a decreased SOFA scores in the L-citrulline group as compared to the placebo group on day 7.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* medical patient (absence of recent surgery or trauma)
* initial aggression < 5 days
* mechanically ventilated with expected duration of mechanical ventilation > 2 days
* exclusive enteral nutrition
* absence of previous immunosuppression

Exclusion Criteria:

* severe sepsis
* septic shock
* obesity defined as BMI above 40
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Organ failure score comparison D7 | At day 7
  Organ failure score (SOFA score) on day 7 in the L-citrulline group as compared to the placebo group

SECONDARY OUTCOMES:
Organ failure score comparison D3 | At day 3
  Organ failure score (SOFA score) on day 3 in the L-citrulline group as compared to the placebo group
SOFA score evolution between randomisation and D7 | up to 7 days
  Binary criterion of success or failure :
  - Success is defined by: an improved SOFA score of at least 2 points from randomization to Day 7 or an improvement in the general condition yielding the release of the unit;
  - Failure is defined by an improved SOFA score but less than 2 points, no improvement or worsening of the SOFA score from randomization to Day 7 or the patient's death before J7;
Expression of HLA-DR | At day 7
  Expression of HLA-DR in the L-citrulline group as compared to the placebo group
Plasmatic concentration of IL6 | At day 7
  Comparison of the plasmatic concentration of interleukin-6 between the L-citrulline group and the placebo group
HLA-DR | At day 7
  Comparison of the percentage of expression of monocytic HLA-DR between the L-citrulline group and the placebo group
Plasmatic concentration of L-arginine | At day 7
  Comparison of the plasmatic concentration of L-arginine and its metabolites between the L-citrulline group and the placebo group
Incidence of nosocomial infections | during the stay in the ICU, an average of 7 days
  Comparison between the L-citrulline group and the placebo group
Length of stay | during the stay in hospital, up to 28 days
  Length of stay in ICU and hospital: Comparison between the L-citrulline group and the placebo group
Mortality | during the stay in hospital, up to 28 days
  * Mortality in intensive care and in hospital : Comparison between the L-citrulline group and the placebo group
  * Duration of mechanical ventilation.
Duration of mechanical ventilation | during the stay in ICU, an average of 7 days
  Duration of mechanical ventilation: Comparison between the L-citrulline group and the placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc TADIE, MD, Principal Investigator — CHU Rennes
Locations (4):
- France (4):
  - CHU Angers, Angers
  - CHU Nantes, Nantes
  - Paris - HEGP, Paris
  - Rennes Hospital University, Rennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tadie JM, Locher C, Maamar A, Reignier J, Asfar P, Commereuc M, Lesouhaitier M, Gregoire M, Le Pabic E, Bendavid C, Moreau C, Diehl JL, Gey A, Tartour E, Le Tulzo Y, Thibault R, Terzi N, Gacouin A, Roussel M, Delclaux C, Tarte K, Cynober L. Enteral citrulline supplementation versus placebo on SOFA score on day 7 in mechanically ventilated critically ill patients: the IMMUNOCITRE randomized clinical trial. Crit Care. 2023 Oct 3;27(1):381. doi: 10.1186/s13054-023-04651-y. PMID 37784110